CLINICAL TRIAL: NCT02946580
Title: A Double-blind, Randomized, Placebo-controlled Trial of Naloxegol for Prevention of Post-operative Constipation in Spinal Surgery Patients
Brief Title: Naloxegol for the Prevention of Constipation in Postoperative Spinal Surgery Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow recruitment and inability to extend funding.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Kyle Staller, MD, MPH, Principle Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2016P001847; ESR-15-11338, D3820L00008 (Other Grant/Funding Number: AstraZeneca)
Record Dates: First submitted 2016-10-17; First posted 2016-10-27 (Estimated); Results first posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-08

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — naloxegol; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MOVANTIK™ (naloxegol) (Experimental): Subjects in the treatment group will be administered MOVANTIK™ (naloxegol) 25 mg tablet or placebo once daily beginning 2 hours after the completion of their surgery until their discharge from the hospital (variable timing). Subjects with renal impairments (creatine clearance rate of less than 60 mL/min) will receive a 12.5 mg dose tablet of naloxegol in place of the 25 mg dose as advised by FDA guidelines. For patients who are unable to swallow the tablet whole, the tablet can be crushed and given orally or administered via nasogastric tube.
  Interventions: Drug: MOVANTIK™ (naloxegol)
- Sugar pill (Placebo Comparator): Matching placebo consists of an inert mixture supplied by AstraZeneca in identical-appearing tablets. Subjects in the placebo group will be administered a placebo tablet once daily beginning 2 hours after the completion of their surgery until their discharge from the hospital (variable timing).
  Interventions: Drug: Sugar Pill

INTERVENTIONS:
Drug: MOVANTIK™ (naloxegol)
  Arms: MOVANTIK™ (naloxegol)
Drug: Sugar Pill
  Arms: Sugar pill

SUMMARY:
Constipation is a known complication of the postoperative period after spinal surgery, where prescription pain medicines called opioids are traditionally used in high doses for the treatment of surgery-related pain. The goal of this study is to determine the effectiveness of Movantik (naloxegol)-a FDA-approved drug used to treat constipation that is caused by opioids-in preventing constipation in patients undergoing spinal fusion surgery at MGH.

DETAILED DESCRIPTION:
We conducted a randomized, double-blind, placebo-controlled trial at a single, academic tertiary center (Massachusetts General Hospital, Boston, MA) from 2017 to 2018. Adult male and female patients between the ages of 18 and 80 who were planned to undergo non-urgent, elective posterior-approach spinal fusion surgeries by the Department of Neurosurgery were eligible for inclusion. Of note, patients with preexisting opioid and/or laxative use were still considered eligible and patients were not stratified according to these characteristics. Once a surgeon and the patient made a joint decision to proceed with elective, posterior spinal fusion surgery, patients would be approached by study personnel, with all eligible patients recruited independently of their surgeon to ensure no conflict of interest. After informed consent, eligible patients provided baseline demographic information including age, sex, race, pre-operative laxative use, and pre-operative opioid use. In addition, subjects completed a Bowel Function Index (BFI), a validated measure of opioid-induced constipation.10 Patients were not instructed to alter their daily regimen from time of consent to initiation of the study. On the day prior to scheduled surgery, clinical research pharmacy staff randomized subjects in a 1:1 ratio. With the exception of the pharmacist preparing the study drug or placebo, who was unaffiliated with the investigators or study sponsor, the individual treatment assignment was unknown to study staff, patients, sponsors, and clinical treatment teams.

Upon completion of surgery, post operative care unit nurses administered 25 mg of oral naloxegol (12.5 mg for creatinine clearance of <60 mL/min) or an identical placebo within 2 hours of arrival in the recovery room post-operatively and then every 24 hours thereafter

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between the ages of 18 and 75 years undergoing non-urgent, elective spinal fusion at Massachusetts General Hospital who are admitted to the neurosurgery floor from the operating room

Exclusion Criteria:

* Patients who are taken to the operating room from another inpatient floor or service (already hospitalized prior to surgery)
* Patients with evidence of bowel obstruction
* Patients unable to take oral medications by mouth or by enteric feeding tube (gastrostomy or jejunostomy)
* Patients with a documented or potential allergy or adverse reaction to Movantik (naloxegol) from outpatient use
* Patients currently taking Movantik (naloxegol) in the outpatient setting
* Patients with a preoperative diagnosis of irritable bowel syndrome (IBS) obtained via Rome III questionnaire on screening
* Patients with disruptions to the blood-brain barrier (eg, multiple sclerosis, recent brain injury, Alzheimer's disease, and uncontrolled epilepsy)
* Patients with a history of cancer.
* Patients concomitantly using strong CYP3A4 inhibitors (eg, clarithromycin, ketoconazole), strong CYP3A4 inducers and other opioid antagonists.
* Patients with severe hepatic impairment.
* Patients with a previous history of or risk of bowel perforation.
* Patients with a post-op regional anesthetic technique employed like a continuous epidural or spinal.
* Patients for which local anesthetics will be placed in the wound.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-01; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Staller, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- MOVANTIK™ (Naloxegol): Subjects in the treatment group will be administered MOVANTIK™ (naloxegol) 25 mg tablet or placebo once daily beginning 2 hours after the completion of their surgery until their discharge from the hospital (variable timing). Subjects with renal impairments (creatine clearance rate of less than 60 mL/min) will receive a 12.5 mg dose tablet of naloxegol in place of the 25 mg dose as advised by FDA guidelines. For patients who are unable to swallow the tablet whole, the tablet can be crushed and given orally or administered via nasogastric tube.
  MOVANTIK™ (naloxegol)
- Sugar Pill: Matching placebo consists of an inert mixture supplied by AstraZeneca in identical-appearing tablets. Subjects in the placebo group will be administered a placebo tablet once daily beginning 2 hours after the completion of their surgery until their discharge from the hospital (variable timing).
  Sugar Pill
Period: Overall Study
Arm/Group | MOVANTIK™ (Naloxegol) | Sugar Pill
Started | 28 | 25
Completed | 27 | 20
Not Completed | 1 | 5
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Adverse Event | 0 | 2
Not completed — Did not undergo posterior spinal fusion | 0 | 1

BASELINE CHARACTERISTICS:
Population: One patient out of the 53 enrolled in our study did not undergo posterior fusion surgery and thus was excluded from our analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | MOVANTIK™ (Naloxegol) | Sugar Pill | Total
Number analyzed (Participants) | 28 | 24 | 52
Age, Categorical [Count of Participants; unit: Participants] — Population: One patient out of the 53 enrolled in our study did not undergo posterior fusion surgery and thus was excluded from our analysis.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 12 | 11 | 23
    >=65 years | 16 | 13 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (9.4) | 64.6 (8.7) | 64.6 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 15 | 11 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 25 | 22 | 47
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 24 | 52

OUTCOME MEASURES:

1. Primary Outcome: Time to First Post-operative Spontaneous Bowel Movement
Description: The primary endpoint of the study was time to first post-operative bowel movement, as defined by the first spontaneous bowel movement reported by nursing staff after transfer from the surgical suite to the inpatient floor. A bowel movement was defined as the spontaneous passage of one tablespoon or more of liquid or solid stool (excluding flatus), which could be measured and verified by nursing staff. Time was measured in hours post-operatively with the starting time point marked at the end of the surgical procedure.
Time Frame: through study completion, an average of 6 days
Measure: Mean (Inter-Quartile Range); unit: hours
Arm/Group | MOVANTIK™ (Naloxegol) | Sugar Pill
Number analyzed (Participants) | 28 | 24
hours | 91 [22 to 186] | 94 [43 to 152]

2. Secondary Outcome: Time to Rescue Laxative Medication Use During Hospitalization
Description: The use of a rescue laxative medication is defined as the administration of an additional bowel medication due to a decision by the clinical treatment team that the subject suffered from constipation and required a "rescue" bowel medication. Of note, this medication did not include the study drug, placebo, or the standing laxative orders used in all patient (docusate and sennosides). By definition, a rescue medication could only be given before a subject's first bowel movement or discharge
Time Frame: upon discharge from hospital, an average of 5 days
Population: Patients who received rescue laxative medication while hospitalized.
Measure: Mean (Full Range); unit: hours
Arm/Group | MOVANTIK™ (Naloxegol) | Sugar Pill
Number analyzed (Participants) | 15 | 10
hours | 70 [17.1 to 183.0] | 75 [46.0 to 96.9]

3. Secondary Outcome: Length of Stay
Time Frame: through study completion, an average of 6 days
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | MOVANTIK™ (Naloxegol) | Sugar Pill
Number analyzed (Participants) | 28 | 24
hours | 106 (44.7) | 133 (31.6)

4. Secondary Outcome: Patient's Satisfaction With Their Bowels by Use of the Bowel Function Index
Description: BFI normal reference range is 0-28.8 (on a scale of 100 for all 3 items summed and divided by 3). Higher scores mean a worse outcome.
Time Frame: through study completion, an average of 6 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MOVANTIK™ (Naloxegol) | Sugar Pill
Number analyzed (Participants) | 28 | 24
score on a scale | 14.3 (19.8) | 16.9 (21.5)

5. Secondary Outcome: Patient's Satisfaction With Their Bowels at Discharge Using a 5-point Likert Scale.
Description: Patients completed a bowel satisfaction questionnaire on day of discharge. 5-point Likert scale, "Very dissatisfied" to "Very satisfied." Higher scores mean a better outcome.
Time Frame: upon discharge from hospital, an average of 5 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MOVANTIK™ (Naloxegol) | Sugar Pill
Number analyzed (Participants) | 28 | 24
score on a scale | 3.4 (1.3) | 3.3 (1.4)

6. Secondary Outcome: Number of Participants That Experienced Diarrhea
Time Frame: through study completion, an average of 6 days
Measure: Count of Participants; unit: Participants
Arm/Group | MOVANTIK™ (Naloxegol) | Sugar Pill
Number analyzed (Participants) | 28 | 24
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data was collected throughout hospitalization and 3 days after discharge, or until first post-operative bowel movement if it occurred >3 days after discharge, up to 2 weeks.
Arm/Group | MOVANTIK™ (Naloxegol) | Sugar Pill
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/28 | 1/24
Other Adverse Events (participants affected / at risk) | 1/28 | 1/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MOVANTIK™ (Naloxegol) (N=28) | Sugar Pill (N=24)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MOVANTIK™ (Naloxegol) (N=28) | Sugar Pill (N=24)
Constipation resulting in re-admission to Emergency Department (Gastrointestinal disorders) | 1 (1) | 0 (0) — Admission to emergency department on day 4 post discharge due to constipation
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-02): https://cdn.clinicaltrials.gov/large-docs/80/NCT02946580/Prot_SAP_000.pdf